CLINICAL TRIAL: NCT00604435
Title: Phase II Trial of Neoadjuvant Recombinant Human Endostatin, Docetaxel and Epirubicin as First-line Therapy in Patients With Breast Cancer
Brief Title: Neoadjuvant Endostatin and Chemotherapy for Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Dai-Ming Fan, Principal of Fourth Military Medical University, Fourth Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Endostar B-01; XOBCR01 (Other Grant/Funding Number: Natural Science Foundation of Shaanxi Province (2008K09-06))
Record Dates: First submitted 2008-01-16; First posted 2008-01-30 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; neoadjuvant chemotherapy; docetaxel; epirubicin; recombinant human endostatin (endostar); chemotherapy; endostatin
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Epirubicin; Endostatins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chemotherapy (Active Comparator): neoadjuvant therapy with 3 cycles of Docetaxel and Epirubicin
  Interventions: Drug: docetaxel and epirubicin
- chemotherapy plus endostatin (Experimental): neoadjuvant therapy with 3 cycles of Docetaxel and Epirubicin plus endostatin
  Interventions: Drug: docetaxel and epirubicin plus endostatin

INTERVENTIONS:
Drug: docetaxel and epirubicin — docetaxel 75mg/m2, IV (in the vein) on day 1 of each 21 day cycle; epirubicin 60 mg/m2, IV (in the vein) on day 1 of each 21 day cycle, totally 3 cycles
  Other Names: docetaxel, Sanofi-Aventis; epirubicin, Pfizer
  Arms: chemotherapy
Drug: docetaxel and epirubicin plus endostatin — docetaxel 75mg/m2, IV (in the vein) on day 1 of each 21 day cycle; epirubicin 60 mg/m2, IV (in the vein) on day 1 of each 21 day cycle; endostatin 7.5mg/m2, IV (in the vein) on 1st to 14th days of each 21 day cycle; every 3 weeks, totally 3 cycles
  Other Names: recombinant human endostatin, Simcere Co. China
  Arms: chemotherapy plus endostatin

SUMMARY:
This study was designed to determine the efficacy and safety of neoadjuvant docetaxel and epirubicin (DE) with or without human recombinant endostatin (endostar) for breast cancer patients. The hypothesis of this protocol is that a combined angiogenesis inhibiting therapy to chemotherapy could further enhance the cytotoxic activity in breast cancer.

DETAILED DESCRIPTION:
This is an open labelled, prospective, randomized, phase II clinical trial. A total of 60 patients with core-biopsy confirmed breast cancer, stage ⅡA to ⅢC, and to be treated with neoadjuvant systemic therapy are eligible for entry into this study. Patients will be allocated randomly to two groups to receive either 3 cycles of neoadjuvant DE and endostar or 3 cycles of neoadjuvant DE. All cases receive mammography, contrast-enhanced ultrasound (CEUS), magnetic resonance angiography (MRA), and positron emission tomography (PET) scanning pre- and post-neoadjuvant therapy, and then undergo surgical resection. The primary endpoint is clinical/pathological response. The secondary endpoint is (1) the safety and tolerability of the regimens, (2) the role of mammography, CEUS, MRA and PET for response evaluation, and (3) angiogenic profile and biological information involved in tumor response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer (core needle biopsy for breast cancer diagnosis and fine needle aspiration for lymph node metastasis diagnosis)
* Stage ⅡA-ⅢC
* Age 18-70
* ECOG performance status 0-2
* No evidence of distant metastasis
* No previous therapy
* Normal hematologic function
* left ventricular ejection fraction greater than 50 percent
* No abnormality of renal or liver function
* Written informed consent

Exclusion Criteria:

* With allergic constitution or possible allergic reflection to drugs to be used in this study
* Any concurrent uncontrolled medical or psychiatric disorder
* History of severe heart diseases, including congestive heart failure, unstable angina, uncontrolled arrhythmia, myocardial infarction, uncontrolled high blood pressure, or heart valve disease.
* History of bleeding diathesis
* Being pregnant or nursing

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2008-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
clinical/pathological response | one year

SECONDARY OUTCOMES:
safety and tolerability | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ling Wang, MD, Study Director — Air Force Military Medical University, China; Jianghao Chen, MD, PhD, Study Chair — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Li J, Dong X, Xu Z, Jiang X, Jiang H, Krissansen GW, Sun X. Endostatin gene therapy enhances the efficacy of paclitaxel to suppress breast cancers and metastases in mice. J Biomed Sci. 2008 Jan;15(1):99-109. doi: 10.1007/s11373-007-9201-3. Epub 2007 Aug 18. PMID 17705027
- [Derived] Chen J, Yao Q, Li D, Zhang J, Wang T, Yu M, Zhou X, Huan Y, Wang J, Wang L. Neoadjuvant rh-endostatin, docetaxel and epirubicin for breast cancer: efficacy and safety in a prospective, randomized, phase II study. BMC Cancer. 2013 May 21;13:248. doi: 10.1186/1471-2407-13-248. PMID 23693018